CLINICAL TRIAL: NCT04818255
Title: Stimulation to Improve Memory: PET Education & Disclosure
Brief Title: STIM+: PET Biomarker Education & Disclosure
Acronym: STIM+
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Benjamin Hampstead, PhD, Professor, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: HUM00188109; R01AG058724 (NIH)
Record Dates: First submitted 2021-03-03; First posted 2021-03-26 (Actual); Results first posted 2026-01-29 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Mild Cognitive Impairment; Dementia; Alzheimer's Type (Etiology)
MeSH Terms: conditions — Cognitive Dysfunction; Dementia

STUDY DESIGN:
Intervention Model Description: Participants and care partners who demonstrate intact decisional capacity to engage in PET biomarker disclosure, and who wish to receive the participant's PET results will be provided with education, results, and recommendations for next steps and supportive resources (the intervention). After this intervention, participants will complete follow-up evaluations of mood and anxiety within one week and at six weeks post disclosure.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Disclosure (Experimental): Participants who demonstrated decisional capacity for and interest in disclosure (or whose care partner is able to do so) will receive the participant's personalized PET amyloid and tau biomarker status, as well as information about the meaning and clinical utility of this information and recommendations for next steps (e.g., discussing findings with his/her provider).
  Interventions: Behavioral: PET Biomarker Disclosure

INTERVENTIONS:
Behavioral: PET Biomarker Disclosure — Participants receive information about whether they currently have elevated or not-elevated amyloid and/or tau based on recent PET imaging conducted as part of an affiliated research study (no additional imaging is required for this project). Participants meet with a licensed clinical neuropsychologist to discuss their biomarker status, the meaning of this information, and potential next steps to consider based of their status. Participants receive written summaries of this information, as well as resources as deemed necessary or as requested.

SUMMARY:
When dementia is caused by AD, we refer to it as dementia of the Alzheimer's Type (DAT). The greatest risk factor for Alzheimer's Disease (AD) and DAT is advancing age, but DAT is not a normal part of aging. Studies have shown that changes in the brain happen before full symptoms of DAT develop. These changes include a buildup of two proteins within the brain, called amyloid and tau. The two goals of this study are

(1) to determine whether patients with mild cognitive impairment or dementia-Alzheimer's type (DAT) are able to demonstrate decisional capacity to engage in PET amyloid and tau disclosure after receiving education; and (2) to assess how patients and care partners react to PET amyloid and tau biomarker disclosure.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in the Stimulation to Improve Memory Study (NCT03875326).
* Completed PET scan with amyloid and/or tau tracer success.
* Demonstrates decision-making capacity to engage in PET disclosure, or has a care partner in attendance that demonstrates decision-making capacity for the participant to engage in disclosure
* If diagnosed with DAT: must have a cognitively intact study partner (i.e., their care partner)
* If diagnosed with MCI: strongly recommended to have a cognitively intact study partner (i.e., their care partner)

Exclusion Criteria:

* Active diagnosis of moderate depression or anxiety without treatment
* Newly diagnosed neurologic disease (since completion of Stimulation to Improve Memory Study activities)

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Actual)
Dates: Start 2020-12-10 (Actual); Primary Completion 2024-11-07 (Actual); Study Completion 2024-11-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ben Hampstead, PhD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan Medical School, Department of Psychiatry, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared with researchers outside of this study.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 161 total individuals were recruited for the study; however, 9 screen failed during the screening and consenting process and were not eligible to begin study activities
Groups:
- Amyloid Positive Participants: Participants with amyloid positivity (amyloid positive, tau positive and amyloid positive, tau negative).
- Amyloid Negative Participants: Participants with negative amyloid results (amyloid negative, tau negative and amyloid negative, tau unknown; no participants had amyloid negative, tau positive results)
- Study Partners of Amyloid Positive Participants: Study partners of participants later found to have amyloid positivity
- Study Partners of Amyloid Negative Participants: Study partners of participants later found to be amyloid negative
Period: Education Session
Arm/Group | Amyloid Positive Participants | Amyloid Negative Participants | Study Partners of Amyloid Positive Participants | Study Partners of Amyloid Negative Participants
Started (Began education session) | 60 | 18 | 59 | 11
Completed | 60 | 18 | 59 | 11
Not Completed | 0 | 0 | 0 | 0
Period: Disclosure Sesions
Arm/Group | Amyloid Positive Participants | Amyloid Negative Participants | Study Partners of Amyloid Positive Participants | Study Partners of Amyloid Negative Participants
Started | 55 | 16 | 55 | 8
Completed | 54 | 16 | 54 | 8
Not Completed | 1 | 0 | 1 | 0
Not completed — Lost to Follow-up | 1 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: 152 total individuals were eligible and enrolled in the study; they are characterized below. Of these, 2 dyads (2 participants and 2 study partners) did not enter the Education Session intervention (1 dyad lost to follow-up before session, 1 dyad declined after further consideration). Therefore, 148 total individuals began and completed the Education Session.
Groups:
- Study Partners of Amyloid Positive Participants: Study partners of participants later found to be amyloid positive
- Total: Total of all reporting groups
Arm/Group | Amyloid Positive Participants | Amyloid Negative Participants | Study Partners of Amyloid Positive Participants | Study Partners of Amyloid Negative Participants | Total
Number analyzed (Participants) | 62 | 18 | 61 | 11 | 152
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Missing age data for 1 study partner
  years
    number analyzed (Participants) | 62 | 18 | 60 | 11 | 151
    (all) | 71.55 (7.07) | 71.94 (7.38) | 67.10 (8.96) | 71.09 (9.03) | 71.64 (7.10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 7 | 37 | 6 | 83
  Male | 29 | 11 | 24 | 5 | 69
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 3 | 3 | 2 | 2 | 10
  White | 59 | 12 | 58 | 6 | 135
  More than one race | 0 | 0 | 0 | 1 | 1
  Unknown or Not Reported | 0 | 3 | 0 | 1 | 4
Education [Mean (Standard Deviation); unit: years] — Population: Education data were missing for 1 participant and 3 study partners
  years
    number analyzed (Participants) | 61 | 18 | 59 | 10 | 148
    (all) | 16.08 (2.54) | 15.89 (3.10) | 16.24 (2.90) | 16.00 (2.49) | 16.04 (2.66)

OUTCOME MEASURES:

1. Primary Outcome: Participant Interest in PET Biomarker Disclosure
Description: Percent of participants surveyed who were interested in receiving their PET biomarker feedback following education, prior to disclosure
Time Frame: Immediately Following Pre-Disclosure Education Session (within one month of enrollment)
Population: Only participants were surveyed on their interest in learning biomarker results. At the time of this outcome measure, neither participants nor study team knew the participants' amyloid status; therefore, this outcome was designed to be measured independent of biomarker status.
Measure: Count of Participants; unit: Participants
Groups:
- Participants Who Completed the Pre-disclosure Educational Session: Participants who completed consent and the pre-disclosure education and decision-making assessment session
Arm/Group | Participants Who Completed the Pre-disclosure Educational Session
Number analyzed (Participants) | 78
Participants | 73

2. Primary Outcome: Percent of Individuals Demonstrating Disclosure Decision-making Capacity
Description: This interactive interview involves an assessment of understanding, appreciation, rationale, and communication of a decision regarding participating or not participating in PET biomarker disclosure. During an education session in which information about PET disclosure is reviewed, participants are asked questions to determine how well they comprehend and appreciated risks and benefits of engaging in PET biomarker disclosure. They are provided with prompts/clarification as needed. Examiners subjectively score each response as correct or incorrect and utilize this information to determine whether participants are demonstrate decisional capacity for PET biomarker disclosure. Results are pass (disclosure decisional capacity intact) or fail (disclosure decisional capacity not intact). Therefore, we will measure the percent of individuals who are able to pass this measure.
Time Frame: Immediately Following Pre-Disclosure Education Session (within one month of enrollment)
Population: Decision-making capacity was only measured in participants (not study partners) for the purpose of this aim. The aim also investigated differences in decision-making capacity for biomarker disclosure based on diagnosis (MCI vs. Dementia). At the time that this outcome was assessed, neither participants nor study team knew the participants' biomarker status. Therefore, decision-making capacity was compared only by participant diagnostic group.
Measure: Count of Participants; unit: Participants
Groups:
- Mild Cognitive Impairment: Participants diagnosed with mild cognitive impairment
- Dementia: Participants diagnosed with dementia presumed to be of the Alzheimer's type
Arm/Group | Mild Cognitive Impairment | Dementia
Number analyzed (Participants) | 32 | 46
Participants | 25 | 10
Statistical Analysis 1: Comparison: Mild Cognitive Impairment vs Dementia; Test type: Superiority; p < .001, Chi-squared; Pearson chi-squared = 24.26

3. Primary Outcome: Effect of Disclosure (Time) and Biomarker Status on Positive and Negative Affect Scale - Short Form (PANAS-SF) Positive Subscale Score
Description: This 10-item subscale asks respondents to rate the extent to which they are experiencing positive (e.g., excited, inspired) emotions on a Likert-style scale ranging from '1 = Very Slightly or Not at All' to '5=Extremely.' Scores range from 10-50, with higher scores indicating higher positive emotions.
Time Frame: Change from Baseline to Immediately following disclosure (within 6 months of baseline), 1-week post-disclosure (within 6.5 months of baseline), and 6-weeks post-disclosure (within 8 months of baseline)
Measure: Mean (Standard Deviation); unit: PANAS Positive subscale score
Groups:
- Amyloid Positive: Participants with amyloid positivity (amyloid positive, tau positive and amyloid positive, tau negative).
- Amyloid Negative: Participants with negative amyloid results (amyloid negative, tau negative and amyloid negative, tau unknown; no participants had amyloid negative, tau positive results)
- Study Partners of Amyloid Positive Participants: Study Partners of Participants found to be amyloid positive
- Study Partners of Amyloid Negative Participants: Study Partners of Participants found to be amyloid negative
Arm/Group | Amyloid Positive | Amyloid Negative | Study Partners of Amyloid Positive Participants | Study Partners of Amyloid Negative Participants
Number analyzed (Participants) | 51 | 16 | 49 | 8
PANAS Positive subscale score
  Baseline | 38.53 (5.78) | 36.19 (7.05) | 39.49 (5.76) | 40.63 (6.39)
  Immediate Post-Disclosure | 35.10 (6.77) | 37.31 (7.13) | 37.61 (6.75) | 41.13 (7.06)
  1-Week Post-Disclosure | 35.31 (8.34) | 36.81 (9.03) | 38.27 (6.87) | 42.25 (5.42)
  6-Week Post-Disclosure | 36.10 (7.43) | 36.50 (10.45) | 38.35 (7.12) | 41.13 (6.03)
Statistical Analysis 1: Comparison: Amyloid Positive vs Amyloid Negative; Test type: Superiority; p = .146, Repeated Measures ANOVA; Examined the effect of disclosure (Time) x Amyloid Status effect to evaluate the impact of disclosure and result on PANAS scores
Statistical Analysis 2: Comparison: Study Partners of Amyloid Positive Participants vs Study Partners of Amyloid Negative Participants; Test type: Superiority; p = .499, Repeated Measures ANOVA; Evaluated the effect of disclosure (Time) x participant Amyloid Status on PANAS Positive subscale scores among study partners

4. Primary Outcome: Effect of Disclosure (Time) and Biomarker Status on Positive and Negative Affect Scale - Short Form (PANAS-SF) Negative Subscale Score
Description: This 10-item subscale asks respondents to rate the extent to which they are experiencing positive negative (e.g., distressed, ashamed) emotions on a Likert-style scale ranging from '1 = Very Slightly or Not at All' to '5=Extremely.' The scores range from 10-50, with higher scores indicating higher negative emotions.
Time Frame: Change from Baseline to Immediately following disclosure (within 6 months of baseline), 1-week post-disclosure, and 6-weeks post-disclosure
Measure: Mean (Standard Deviation); unit: PANAS Negative Subscale Score
Arm/Group | Amyloid Positive | Amyloid Negative | Study Partners of Amyloid Positive Participants | Study Partners of Amyloid Negative Participants
Number analyzed (Participants) | 51 | 16 | 49 | 8
PANAS Negative Subscale Score
  Pre-Disclosure | 15.10 (5.16) | 13.31 (4.95) | 15.47 (4.92) | 16.88 (9.60)
  Immediately Post-Disclosure | 14.71 (5.33) | 14.50 (3.92) | 14.73 (3.97) | 16.38 (5.55)
  1-Week Post-Disclosure | 16.22 (6.87) | 13.31 (3.54) | 14.86 (4.70) | 14.75 (4.62)
  6-Week Post-Disclosure | 15.08 (5.23) | 14.56 (4.75) | 14.90 (5.06) | 15.63 (6.93)
Statistical Analysis 1: Comparison: Amyloid Positive vs Amyloid Negative; Test type: Superiority; p = .094, Repeated Measures ANOVA; [statistical method as in outcome 3, analysis 1]
Statistical Analysis 2: Comparison: Study Partners of Amyloid Positive Participants vs Study Partners of Amyloid Negative Participants; Test type: Superiority; p = .476, Repeated Measures ANOVA; Evaluated the effect of disclosure (time) x participant amyloid status on study partners' PANAS negative subscale scores

5. Primary Outcome: Effect of Biomarker Status on Impact of Neuroimaging in Alzheimer's Disease (INI-AD) Distress Score
Description: Measures negative reactions to AD-related personal neuroimaging results received as part of disclosure (0-55; higher scores indicate higher distress) starting from immediately following disclosure to six weeks post-disclosure.
Time Frame: Immediately following disclosure (within 6 months of baseline) to 1-week post-disclosure (within 6.5 months of baseline), and 6-weeks post-disclosure (within 8 months of baseline)
Measure: Mean (Standard Deviation); unit: INI-AD Distress Subscale Total Score
Arm/Group | Amyloid Positive Participants | Amyloid Negative Participants | Study Partners of Amyloid Positive Participants | Study Partners of Amyloid Negative Participants
Number analyzed (Participants) | 52 | 15 | 51 | 8
INI-AD Distress Subscale Total Score
  Immediately Post-Disclosure | 12.15 (10.01) | 1.87 (2.23) | 11.84 (7.42) | 1.50 (2.50)
  1-Week Post-Disclosure | 11.90 (10.62) | 2.47 (5.21) | 11.86 (6.59) | 4.13 (4.52)
  6-Weeks Post-Disclosure | 10.44 (9.09) | 1.93 (3.11) | 12.06 (6.60) | 3.50 (5.21)
Statistical Analysis 1: Comparison: Amyloid Positive Participants vs Amyloid Negative Participants; Test type: Superiority; p < .001, Repeated Measures ANOVA; Examined the between-subjects effect of participant amyloid status on INI-AD Distress subscale score
Statistical Analysis 2: Comparison: Study Partners of Amyloid Positive Participants vs Study Partners of Amyloid Negative Participants; Test type: Superiority; p < .001, Repeated Measures ANOVA; Examined the between-subjects effect of participant amyloid status on study partner INI-AD Distress subscale score

6. Primary Outcome: Effect of Biomarker Status on Impact of Neuroimaging in Alzheimer's Disease (INI-AD) Positive Emotions Score
Description: Measures change in positive reactions to AD-related personal neuroimaging results received as part of disclosure (0-20; higher scores indicate higher positive emotions) starting from immediately following disclosure to six weeks post-disclosure.
Time Frame: as for outcome 5
Measure: Mean (Standard Deviation); unit: INI-AD Positive Subscale Total Score
Arm/Group | Amyloid Positive Participants | Amyloid Negative Participants | Study Partners of Amyloid Positive Participants | Study Partners of Amyloid Negative Participants
Number analyzed (Participants) | 52 | 15 | 51 | 8
INI-AD Positive Subscale Total Score
  Immediately Post-Disclosure | 12.17 (3.47) | 17.93 (3.77) | 11.27 (3.78) | 19.00 (2.14)
  1-Week Post-Disclosure | 10.87 (4.14) | 17.40 (3.33) | 10.82 (3.01) | 18.50 (1.77)
  6-Weeks Post-Disclosure | 11.04 (12.25) | 3.53 (4.57) | 10.25 (2.46) | 17.75 (3.11)
Statistical Analysis 1: Comparison: Amyloid Positive Participants vs Amyloid Negative Participants; Test type: Superiority; p < .001, Repeated Measures ANOVA; Examined the effect of participant amyloid status on participant INI-AD Positive Subscale Scores
Statistical Analysis 2: Comparison: Study Partners of Amyloid Positive Participants vs Study Partners of Amyloid Negative Participants; Test type: Superiority; p < .001, Repeated Measures ANOVA; Evaluated the effect of participant amyloid status on study partner INI-AD Positive Emotions subscale scores

7. Primary Outcome: Effect of Disclosure (Time) and Biomarker Status on Stigma Scale for Chronic Illness (SSCI-8) Total Score
Description: The Stigma Scale for Chronic Illness (SSCI-8) measures perceived and experienced stigma based on a chronic illness (in this case, cognitive disorder). The SSCI-8 demonstrates strong reliability for the measurement of both internalized (perceived) and enacted (experienced) stigma perceived by individuals with chronic neurological conditions. Respondents complete 8 items about experiences of stigma, rated on a Likert-style scale from 1 = 'Never' to 5 = 'Always'. Items are summed to a total score (min=8, max=40) with higher scores suggesting more stigma.
Time Frame: as for outcome 4
Measure: Mean (Standard Deviation); unit: SSCI-8 Total Score
Arm/Group | Amyloid Positive | Amyloid Negative
Number analyzed (Participants) | 50 | 16
SSCI-8 Total Score
  Baseline (Pre-Disclosure) | 11.14 (2.86) | 9.63 (2.06)
  Immediately Post-Disclosure | 9.86 (2.20) | 10.31 (2.75)
  1-Week Post-Disclosure | 10.50 (2.89) | 9.56 (1.90)
  6-Weeks Post-Disclosure | 10.02 (2.77) | 9.69 (2.33)
Statistical Analysis 1: Comparison: Amyloid Positive vs Amyloid Negative; Test type: Superiority; p = .051, Repeated Measures ANOVA; Examined the effect of disclosure (time) by biomarker status on SSCI scores; Mean Difference (Final Values) = 2.68

8. Primary Outcome: Effect of Disclosure (Time) and Biomarker Status on Self-Efficacy for Managing Chronic Disease Scale (SECD) Total Score
Description: The Self-Efficacy for Managing Chronic Disease (SECD) scale is a 6-item scale that measures perceived ability to self-manage the physical, emotional, and cognitive symptoms associated with their chronic disease. Items are listed on a 10-point scale ranging from 1 = 'Not at all confident' to 10 = 'Totally confident'. Item scores are summed and averaged. Lower scores suggest lower confidence in managing symptoms. Higher scores suggest higher confidence in managing symptoms. There are no clinical cut-offs for this measure.
Time Frame: as for outcome 4
Measure: Mean (Standard Deviation); unit: SECD Total Score
Arm/Group | Amyloid Positive | Amyloid Negative
Number analyzed (Participants) | 51 | 16
SECD Total Score
  Baseline (Pre-Disclosure) | 7.96 (1.73) | 8.10 (1.24)
  Immediately Post-Disclosure | 7.94 (1.47) | 8.21 (1.39)
  1-Week Post-Disclosure | 7.32 (2.11) | 8.32 (2.22)
  6-Week Post-Disclosure | 7.48 (1.90) | 8.06 (1.79)
Statistical Analysis 1: Comparison: Amyloid Positive vs Amyloid Negative; Test type: Superiority; p = .399, Repeated Measures ANOVA; Examined the effect of disclosure (time) by biomarker result on SECD Scores; Mean Difference (Final Values) = 0.977

9. Primary Outcome: Effect of Disclosure (Time) and Biomarker Status on Future Time Perspectives Scale (FTP) Average Score
Description: The Future Time Perspective (FTP) scale is a 10-item scale that measures the extent to which respondents feel that they have potential for productive and functional years ahead of them. Statements regarding positive and negative future time perspective are rated on a 7-point Likert-style scale, ranging from 1= 'Very untrue' to 7='Very true.' 3 items are reverse scored, then all items are summed and averaged. Minimum average score is 1, maximum average score is 7. Higher scores suggest greater time perspective.
Time Frame: as for outcome 4
Measure: Mean (Standard Deviation); unit: FTP Total Score
Groups:
- Study Partners of Amyloid Negative Participants: Study Partners of participants founds to be amyloid negative
Arm/Group | Amyloid Positive Participants | Amyloid Negative Participants | Study Partners of Amyloid Positive Participants | Study Partners of Amyloid Negative Participants
Number analyzed (Participants) | 51 | 16 | 49 | 8
FTP Total Score
  Baseline (Pre-Disclosure) | 4.33 (1.10) | 5.00 (0.86) | 4.68 (1.11) | 5.24 (0.76)
  Immediately Post-Disclosure | 4.42 (1.13) | 4.91 (1.03) | 4.56 (1.14) | 5.20 (1.06)
  1-Week Post-Disclosure | 4.35 (1.29) | 4.77 (1.12) | 4.52 (1.03) | 5.20 (1.07)
  6-Weeks Post-Disclosure | 4.23 (1.22) | 4.52 (1.08) | 4.40 (1.00) | 5.09 (1.00)
Statistical Analysis 1: Comparison: Amyloid Positive Participants vs Amyloid Negative Participants; Test type: Superiority; p = .615, Repeated Measures ANOVA; Examined the effect of disclosure (time) by participant amyloid status on FTP scores
Statistical Analysis 2: Comparison: Study Partners of Amyloid Positive Participants vs Study Partners of Amyloid Negative Participants; Test type: Superiority; p = .956, Repeated Measures ANOVA; Evaluated the effect of disclosure (time) x participant amyloid status on study partners' FTP subscale scores

10. Primary Outcome: Effect of Diagnosis on Participant Comprehension/Recall of Results Percent Correct Score: Immediately Following Disclosure
Description: This tool, created for the purpose of this study, measures participant's ability to understand their biomarker results and their meaning. Scores on the nine items are converted into a percent correct score, with higher scores indicating better comprehension and memory of results.
Time Frame: Immediately following disclosure (within 6 months of baseline)
Measure: Mean (Standard Deviation); unit: % correct on comprehension measure
Groups:
- Participants With Mild Cognitive Impairment: Participants diagnosed with mild cognitive impairment
- Participants With Dementia: Participants diagnosed with dementia presumed to be of the Alzheimer's type
- Study Partners of Participants With MCI: Study Partners of participants diagnosed with MCI
- Study Partners of Participants With Dementia: Study partners of participants diagnosed with dementia
Arm/Group | Participants With Mild Cognitive Impairment | Participants With Dementia | Study Partners of Participants With MCI | Study Partners of Participants With Dementia
Number analyzed (Participants) | 28 | 39 | 19 | 37
% correct on comprehension measure | 93.25 (16.09) | 72.27 (23.92) | 98.26 (5.52) | 94.95 (16.17)
Statistical Analysis 1: Comparison: Participants With Mild Cognitive Impairment vs Participants With Dementia; Test type: Superiority; p < .001, t-test, 2 sided
Statistical Analysis 2: Comparison: Study Partners of Participants With MCI vs Study Partners of Participants With Dementia; Test type: Superiority; p = .255, t-test, 2 sided

11. Primary Outcome: Effect of Diagnosis on Participant Comprehension/Recall of Results Percent Correct Score: 1-Week Post-Disclosure
Description: as for outcome 10
Time Frame: 1-week post-disclosure (within 6.5 months of baseline)
Measure: Mean (Standard Deviation); unit: Percent Correct
Arm/Group | Participants With Mild Cognitive Impairment | Participants With Dementia | Study Partners of Participants With MCI | Study Partners of Participants With Dementia
Number analyzed (Participants) | 29 | 41 | 20 | 41
Percent Correct | 86.38 (21.25) | 64.22 (30.30) | 98.80 (3.71) | 98.39 (5.80)
Statistical Analysis 1: Comparison: Participants With Mild Cognitive Impairment vs Participants With Dementia; Test type: Superiority; p < .001, t-test, 2 sided
Statistical Analysis 2: Comparison: Study Partners of Participants With MCI vs Study Partners of Participants With Dementia; Test type: Superiority; p = .740, t-test, 2 sided

12. Primary Outcome: Effect of Diagnosis on Participant Comprehension/Recall of Results Percent Correct Score: 6-Week Post-Disclosure
Description: as for outcome 10
Time Frame: 6 weeks post-disclosure (within 8 months of baseline)
Measure: Mean (Standard Deviation); unit: Percent Correct
Arm/Group | Participants With Mild Cognitive Impairment | Participants With Dementia | Study Partners of Participants With MCI | Study Partners of Participants With Dementia
Number analyzed (Participants) | 29 | 39 | 20 | 39
Percent Correct | 87.79 (18.06) | 62.47 (29.10) | 98.90 (4.92) | 96.77 (8.77)
Statistical Analysis 1: Comparison: Participants With Mild Cognitive Impairment vs Participants With Dementia; Test type: Superiority; p < .001, t-test, 2 sided
Statistical Analysis 2: Comparison: Study Partners of Participants With MCI vs Study Partners of Participants With Dementia; Test type: Superiority; p = .237, t-test, 2 sided

13. Primary Outcome: Preparedness for Caregiving Scale (PCS)
Description: This 8-item measure assesses the degree to which care partners of persons with cognitive impairment (e.g., MCI, DAT) perceive they are prepared for and able to manage various domains of caregiving such as providing physical care and emotional support, setting up in-home support services, and coping with stress due to caregiving. Items use a 5-point likert scale ranging from 0 = 'Not at all prepared' to 4 'Very well prepared'. An average score is generated (min=0, max=4) with higher scores indicating greater preparedness.
Time Frame: Measured at baseline, immediately post-disclosure (within 6 months of baseline), and at 1- (within 6.5 months of baseline) and 6-weeks post-disclosure (within 8 months of baseline)
Measure: Mean (Standard Deviation); unit: PCS total score
Arm/Group | Study Partners of Amyloid Positive Participants | Study Partners of Amyloid Negative Participants
Number analyzed (Participants) | 47 | 8
PCS total score
  Baseline | 2.95 (0.62) | 3.52 (0.49)
  Immediately Post-Disclosure | 3.06 (0.58) | 3.66 (0.45)
  1-Week Post-Disclosure | 3.07 (0.66) | 3.53 (0.53)
  6-Weeks Post-Disclosure | 3.01 (0.69) | 3.51 (0.58)
Statistical Analysis 1: Comparison: Study Partners of Amyloid Positive Participants vs Study Partners of Amyloid Negative Participants; Test type: Superiority; p = .835, Repeated Measures ANOVA; Evaluated the effect of disclosure (time) by participant amyloid status on study partner PCS scores

14. Primary Outcome: Revised Scale for Caregiving Self-Efficacy
Description: The Revised Scale for Caregiving Self-Efficacy is a 15-item scale consisting of 3 sub-scales, each containing 5-items, designed to measure perceived ability to manage aspects related to caregiving among caregivers of persons with dementia. Only one subscale was administered in this study: this 5-item subscale is used to measure the co-participant's perceived ability to manage the emotional stresses associated with caregiving. This measure will be administered to study partners only. Items are averaged (min=0, max=100) with higher scores indicating greater perceived confidence to manage the emotional stressed of caregiving.
Time Frame: as for outcome 13
Measure: Mean (Standard Deviation); unit: total subscale score
Arm/Group | Study Partners of Amyloid Positive Participants | Study Partners of Amyloid Negative Participants
Number analyzed (Participants) | 47 | 8
total subscale score
  Baseline | 81.69 (13.62) | 83.88 (15.01)
  Immediately Post-Disclosure | 80.55 (14.25) | 94.88 (5.25)
  1-Week Post-Disclosure | 81.26 (14.44) | 86.10 (10.50)
  6-Weeks Post-Disclosure | 77.76 (15.59) | 88.83 (7.93)
Statistical Analysis 1: Comparison: Study Partners of Amyloid Positive Participants vs Study Partners of Amyloid Negative Participants; Test type: Superiority; p = .037, Repeated Measures ANOVA; Evaluated the effect of disclosure (time) x participant amyloid status on study partner RSSE scores

ADVERSE EVENTS:
Time Frame: From enrollment until the end of follow-up, up to 9 months
Groups:
- Study Partners of Amyloid Positive Participants: Study partners of amyloid positive participants
- Study Partners of Amyloid Negative Participants: Study partners of amyloid negative participants
Arm/Group | Amyloid Positive Participants | Amyloid Negative Participants | Study Partners of Amyloid Positive Participants | Study Partners of Amyloid Negative Participants
All-Cause Mortality (participants affected / at risk) | 0/60 | 0/18 | 0/59 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/60 | 0/18 | 0/59 | 0/11
Other Adverse Events (participants affected / at risk) | 0/60 | 0/18 | 0/59 | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (5):
  • Study Protocol and Statistical Analysis Plan (2025-06-23): https://cdn.clinicaltrials.gov/large-docs/55/NCT04818255/Prot_SAP_004.pdf
  • Informed Consent Form: Participant Consent - Education (2022-09-08): https://cdn.clinicaltrials.gov/large-docs/55/NCT04818255/ICF_000.pdf
  • Informed Consent Form: Participant Consent - Disclosure (2022-09-08): https://cdn.clinicaltrials.gov/large-docs/55/NCT04818255/ICF_001.pdf
  • Informed Consent Form: Co-Participant Consent - Education (2022-09-08): https://cdn.clinicaltrials.gov/large-docs/55/NCT04818255/ICF_002.pdf
  • Informed Consent Form: Co-Participant Consent - Disclosure (2022-09-08): https://cdn.clinicaltrials.gov/large-docs/55/NCT04818255/ICF_003.pdf